CLINICAL TRIAL: NCT00081744
Title: A Multicenter, Double-Blind, Randomized Comparison Study Of the Efficacy and Safety of Tigecycline to Imipenem/ Cilastatin to Treat Complicated Intra-Abdominal Infections in Hospitalized Subjects
Brief Title: Study Comparing Tigecycline to Imipenem/Cilastatin in Complicated Intra-Abdominal Infections in Hospitalized Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 3074A1-301
Record Dates: First submitted 2004-04-19; First posted 2004-04-21 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Gram-Positive Bacterial Infections; Cross Infection
Keywords: Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Cross Infection; Bacterial Infections | interventions — Tigecycline

INTERVENTIONS:
Drug: Tigecycline

SUMMARY:
Purpose: To provide a mechanism for the emergency use of tigecycline in the appropriate clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≥ 8 years of age and a weight of ≥ 35 kilograms
* Subjects with selected culture-positive infections caused by a multiple antibiotic-resistant pathogen presumed to be susceptible to tigecycline
* Subjects who have failed or are intolerant of other available appropriate antibiotic therapies or whose pathogens are resistant to other available antibiotics

Exclusion Criteria:

* Subjects who are moribund with an expected survival of less than 2 weeks.
* Subjects who have been designated as "Do Not Resuscitate", unless it is anticipated within a reasonable degree of medical certainty that they can achieve benefit from potentially curative antibiotic therapy
* Known or suspected hypersensitivity to tigecycline, tetracyclines, or other compounds related to this class of antibacterial agents

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2002-11; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Result] Oliva ME, Rekha A, Yellin A, Pasternak J, Campos M, Rose GM, Babinchak T, Ellis-Grosse EJ, Loh E; 301 Study Group. A multicenter trial of the efficacy and safety of tigecycline versus imipenem/cilastatin in patients with complicated intra-abdominal infections [Study ID Numbers: 3074A1-301-WW; ClinicalTrials.gov Identifier: NCT00081744]. BMC Infect Dis. 2005 Oct 19;5:88. doi: 10.1186/1471-2334-5-88. PMID 16236177
- [Derived] Fomin P, Koalov S, Cooper A, Babinchak T, Dartois N, De Vane N, Castaing N, Tellado J; 301 And 306 Study Groups. The efficacy and safety of tigecycline for the treatment of complicated intra-abdominal infections - the European experience. J Chemother. 2008 Oct;20 Suppl 1:12-9. doi: 10.1179/joc.2008.20.Supplement-1.12. PMID 19036670